CLINICAL TRIAL: NCT02416297
Title: Three- Dimensional Evaluation of Accelerated Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LIANA FATTORI ABATI (Other)
Responsible Party: Sponsor-Investigator, LIANA FATTORI ABATI, Master degree student, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fattori-001
Record Dates: First submitted 2015-03-27; First posted 2015-04-15 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Malocclusion
Keywords: malocclusion; accelerated tooth movement; Tomography; Extraction
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micro-osteoperforation (Experimental): Minimally invasive micro-osteoperforation procedure used to achieve accelerated orthodontic tooth movement. Topical and local anesthetic will be delivered in the area to be treated in accordance with standard practice.
  Interventions: Procedure: Micro-osteoperforation
- Control (No Intervention): Anterior retraction after premolars extraction will be done conventionally (slide mechanics)

INTERVENTIONS:
Procedure: Micro-osteoperforation — Flapless cortical perforations will be made 8 months minimum after dental extraction. Surgical protocol will be flapless to preserve periodontal health. After local anesthesia, 3 micro osteoperforations will be done with manual instrument, between apex to the contour of free gum between the canine and second pre-molar. Perforations near each tooth will have 6-8 mm depth
  Arms: Micro-osteoperforation

SUMMARY:
The purpose of this research study is to assess the clinical effectiveness of a minimally invasive alveolar microperforation procedure to achieve accelerated tooth movement in patients undergoing orthodontic treatment for orthognathic surgery. "Accelerated tooth movement" means that Microperforation technique may help complete orthodontic treatment sooner than would be expected in conventional orthodontic treatment

DETAILED DESCRIPTION:
SAMPLE: For this prospective study, 22 subjects were selected, with skeletal discrepancies randomly divided into two groups: 1 - accelerated tooth movement technique (ATMT) and 2 - Control .

METHODS: MATERIAL - Orthodontic records done in two times, initial and preoperative; Plaster models of dental extracted jaw every 28 days converted in digital models; Cone Beam Computed tomography done in two times, initial and in the end of extraction space closure.

METHODS: Pre-molar extraction was performed before the Orthodontic Treatment to eliminate the RAP from the tooth extraction. After, at minimum 8 months for leveling, the extraction space closure was activated with light orthodontic traction (200 g each side) in anterior teeth, to maintain therapeutic osteopenia until contact point between the canine the second pre-molar is reached. Slide mechanic was chosen to performed anterior retraction on TADs in IZC.

Cortical perforations - ATMT Group: Flapless cortical micro-osteoperforations has been performed in the dental extraction area. Surgical protocol is flapless to preserve periodontal health. After local anesthesia, 3 micro osteoperforations are done with manual instrument, between the contour of free gum and tooth apex, and the canine and second pre-molar roots. The perforations near each tooth adjacent to the extraction area has 6-8 mm depth.

Results: On digital models - shortest distance between two adjacent teeth to the extraction space will be measured until the space closure.

Cone-Beam Computed Tomography: after image acquisition , data will be previously converted to DICOM , to converted to GIPL in ITK-SNAP 3.2 software. In Slicer software voxels will be converted to size 0.5 mm for further construction of virtual three-dimensional models, through segmentation of anatomical structures again in ITK-SNAP 3.2 software. This segmentation will be made by the full selection of all maxilla and mandible anatomically and individually, with the limit all skeletal outline available, including teeth. After 3D models generation, specific control targeting to fill all narrow spaces, so that they are not excluded from the virtual model and the external cortical displacements are the only ones to be computed in the comparative evaluation between later time. Then regional overlay 3D models will be done using Slicer software. For overlapping structures: In mandible will use along the edge of the mandibular symphysis; maxilla, posterior nasal spine. Overlap is automatic because software compares voxels grayscale to reference region to overlap spatially. Displacement evaluation will be done with Slicer software through colorful maps generated by calculating the distances between points of two representatives surfaces. These maps differentiate the movements between surfaces. For quantification metric, specific online tool is used to measure the displacement in millimeters. We will evaluate quantitative displacement for space closure, closing speed, the possible changes throughout the maxillomandibular complex and compared between groups. After collecting data, the results will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 18-35 years old, in good general health, with adult complete dentition, regardless of presence of third molars.
* Indication for orthognathic surgery
* Tooth extraction indication for orthodontic treatment
* Do not smoke
* Periodontal and teeth healthy
* Do not use bisphosphonates or corticosteroids

Exclusion Criteria:

* Surgically assisted rapid palatal expansion indication
* cleft lip and palate
* craniofacial syndrome
* mental disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of velocity rate of anterior retraction in conventional mechanics and accelerated tooth movement technique | 6 months
  The micro osteoperforations accelerates tooth moviment - Null hipothesis

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Neto, PhD, Study Chair — University of Sao Paulo; Lucia H Cevidanes, PhD, Study Chair — University of Michigan
Locations (1):
- FOUSP, São Paulo, Brazil